CLINICAL TRIAL: NCT05235971
Title: Behavioral Economic Treatment to Enhance Rural Living
Brief Title: Behavioral Economic Treatment to Enhance Rural (BETTER) Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lara Coughlin, Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00181940; 1K23AA028232 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use, Unspecified
Keywords: Heavy alcohol consumption; Alcohol misuse
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Episodic Future thinking (EFT) (Experimental): Participants will receive up to 3 messages a day that include assessment and intervention messages.The messages will describe positive, non-alcohol related events at future time points to facilitate extension of temporal consideration toward future-focused perspectives.
  Interventions: Behavioral: Episodic Future thinking
- Volitional choice (VC) (Experimental): VC creates structured if-then plans to dismantle context-linked alcohol use. Participants will receive up to 3 messages a day that include assessment and intervention messages.
  Interventions: Behavioral: Volitional choice
- Episodic Future thinking plus Volitional choice (Experimental): Participants will receive both EFT and VC interventions with text messages.
  Interventions: Behavioral: Episodic Future thinking; Behavioral: Volitional choice
- Monitoring only (Other): This is a control group in which participants will receive general psychoeducation.
  Interventions: Behavioral: Monitoring only

INTERVENTIONS:
Behavioral: Episodic Future thinking — During a visit with the study team, participants will identify personally-relevant reminders, or cues, that they will receive up to 3 messages a day via text-message over a two-week period.
  The messages will describe positive, non-alcohol related events at future time points to facilitate extension of temporal consideration toward future-focused perspectives.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected
  Arms: Episodic Future thinking (EFT); Episodic Future thinking plus Volitional choice
Behavioral: Volitional choice — Volitional choice creates structured if-then plans to dismantle context-linked alcohol use The messages sent over a two-week period facilitate alternative, healthier choices by identifying and linking risky cues with alternative actions. Participants will receive up to 3 messages a day for 14 days that include assessment and intervention messages.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected.
  Arms: Episodic Future thinking plus Volitional choice; Volitional choice (VC)
Behavioral: Monitoring only — Participants will receive general psychoeducation about alcohol use, mental health, resources, and a description of the assessments to be completed over a two-week field testing period.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected.
  Arms: Monitoring only

SUMMARY:
The purpose of this trial is to get feedback to help develop programs delivered by phone and text messages to improve wellness and health behaviors. This study will enroll adult participants that have been seen in primary care settings and live in rurally designated areas.

DETAILED DESCRIPTION:
This study will evaluate acceptability and feasibility of two remotely-delivered behavioral economic intervention components, alone and in combination, using remote text message delivery. The two intervention components are an episodic future thinking component and a volitional choice component. The goal of this work is to develop and determine acceptability and feasibility of a well-specified, accessible, and theory-driven mobile health intervention to reduce harmful alcohol use in people living in rural regions.

ELIGIBILITY:
Screening Inclusion Criteria:

* adults presenting in Michigan Medicine primary care
* home address in a rurally designated area (e.g., zip code, county),
* documented alcohol use in the Electronic Health Record (EHR) (e.g., alcohol use disorder diagnosis, alcohol misuse or heavy alcohol consumption).

Baseline inclusion criteria:

* an Alcohol Use Disorders Identification Test (AUDIT-C) score of ≥3 in females or ≥4 in males
* regular access to an internet-enabled device (e.g., smart phone, computer, tablet).

Exclusion Criteria:

* Does not understand English
* currently pregnant
* unable to provide informed consent due to medical/psychiatric reasons
* currently in treatment for a substance use disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Coughlin, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hellman L, Wilkins C, Bayrakdarian N, Jannausch M, Bonar EE, Walton MA, Lin LA, Staton M, Coughlin L. Rural- and nonrural-specific themes in personalized intervention messages for adults with at-risk alcohol use living in rural areas. Exp Clin Psychopharmacol. 2026 Feb;34(1):8-17. doi: 10.1037/pha0000830. PMID 41538227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a large tertiary healthcare system from May 2022 through April 2023.
Groups:
- Episodic Future Thinking (EFT): Participants will receive up to 3 messages a day that include assessment and intervention messages.The messages will describe positive, non-alcohol related events at future time points to facilitate extension of temporal consideration toward future-focused perspectives.
  Episodic Future thinking: During a visit with the study team, participants will identify personally-relevant reminders, or cues, that they will receive up to 3 messages a day via text-message over a two-week period.
  The messages will describe positive, non-alcohol related events at future time points to facilitate extension of temporal consideration toward future-focused perspectives.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected
- Volitional Choice (VC): VC creates structured if-then plans to dismantle context-linked alcohol use. Participants will receive up to 3 messages a day that include assessment and intervention messages.
  Volitional choice: Volitional choice creates structured if-then plans to dismantle context-linked alcohol use The messages sent over a two-week period facilitate alternative, healthier choices by identifying and linking risky cues with alternative actions. Participants will receive up to 3 messages a day for 14 days that include assessment and intervention messages.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected.
- Episodic Future Thinking Plus Volitional Choice: Participants will receive both EFT and VC interventions with text messages.
  Episodic Future thinking: During a visit with the study team, participants will identify personally-relevant reminders, or cues, that they will receive up to 3 messages a day via text-message over a two-week period.
  The messages will describe positive, non-alcohol related events at future time points to facilitate extension of temporal consideration toward future-focused perspectives.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected
  Volitional choice: Volitional choice creates structured if-then plans to dismantle context-linked alcohol use The messages sent over a two-week period facilitate alternative, healthier choices by identifying and linking risky cues with alternative actions. Participants will receive up to 3 messages a day for 14 days that include assessment and intervention messages.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected.
- Monitoring Only: This is a control group in which participants will receive general psychoeducation.
  Monitoring only: Participants will receive general psychoeducation about alcohol use, mental health, resources, and a description of the assessments to be completed over a two-week field testing period.
  In addition, participants will have phone meetings (video or not) where health behaviors as well as survey information is noted and collected.
Period: Overall Study
Arm/Group | Episodic Future Thinking (EFT) | Volitional Choice (VC) | Episodic Future Thinking Plus Volitional Choice | Monitoring Only
Started | 17 | 21 | 19 | 18
Completed | 17 | 21 | 19 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Episodic Future Thinking (EFT) | Volitional Choice (VC) | Episodic Future Thinking Plus Volitional Choice | Monitoring Only | Total
Number analyzed (Participants) | 17 | 21 | 19 | 18 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 13 | 12 | 54
  >=65 years | 5 | 4 | 6 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (19.8) | 54.7 (13.4) | 58.0 (14.8) | 53.9 (16.5) | 55.2 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 12 | 12 | 47
  Male | 7 | 8 | 7 | 6 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian/Alaskan Native | 0 | 0 | 0 | 0 | 0
  Race/Ethnicity: Asian | 0 | 0 | 0 | 0 | 0
  Race/Ethnicity: Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race/Ethnicity: Black/African American | 0 | 0 | 0 | 0 | 0
  Race/Ethnicity: White | 17 | 21 | 19 | 17 | 74
  Race/Ethnicity: More than one race | 0 | 0 | 0 | 1 | 1
  Race/Ethnicity: Don't know/Refuse | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 21 | 19 | 18 | 75
Alcohol Use Severity (AUDIT) [Mean (Standard Deviation); unit: scores on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviors, and alcohol-related problems. The AUDIT ranges from a score of 0 to 40 with higher values indicating riskier drinking and lower values indicating lower risk.
  Total scores of 8 or more are recommended as indicators of hazardous and harmful alcohol use, including possible alcohol dependence. The total AUDIT score will reflect the patient's level of risk related to alcohol.
  scores on a scale | 7.2 (5.7) | 7.5 (6.8) | 8.4 (8.0) | 8.6 (6.8) | 7.9 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Intervention - Screening
Description: Percent of participants who complete intervention phone call
Time Frame: Day 1 of Intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Episodic Future Thinking (EFT) | Volitional Choice (VC) | Episodic Future Thinking Plus Volitional Choice | Monitoring Only
Number analyzed (Participants) | 17 | 21 | 19 | 18
Participants | 17 | 21 | 19 | 18

2. Primary Outcome: Feasibility of the Intervention - Enrollment
Description: Percent of participants who elect to receive text messages
Time Frame: Day 1 of Intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Episodic Future Thinking (EFT) | Volitional Choice (VC) | Episodic Future Thinking Plus Volitional Choice | Monitoring Only
Number analyzed (Participants) | 17 | 21 | 19 | 18
Participants | 17 | 21 | 19 | 18

3. Primary Outcome: Intervention Acceptability: Number of Participants Who Rated the Intervention as Acceptable
Description: Number of participants with positive acceptability ratings who indicated enjoying the intervention at least a little bit. In a phone survey, participants were asked to rate their enjoyment of the intervention on a scale of 1-5, where 1 was "not at all" and 5 was "extremely". Scores of 2 ("a little bit") or more were considered to be positive indicators of acceptability.
Time Frame: 2 Weeks Post-Intervention
Population: This measure is reported among all intervention groups and the control group to determine their level of enjoyment with participating in the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Episodic Future Thinking (EFT) | Volitional Choice (VC) | Episodic Future Thinking Plus Volitional Choice | Monitoring Only
Number analyzed (Participants) | 17 | 21 | 19 | 18
Participants | 17 | 19 | 19 | 17

4. Secondary Outcome: Alcohol Consumption
Description: Average number of standard drinks consumed during the 2-week intervention period per person. A "standard drink" was considered to be 12 oz beer, 1.5 ounce shot of liquor, or 5 oz glass of wine.
Time Frame: The 2 weeks (14-days) of the intervention period
Measure: Mean (Standard Deviation); unit: standard drinks per person
Arm/Group | Episodic Future Thinking (EFT) | Volitional Choice (VC) | Episodic Future Thinking Plus Volitional Choice | Monitoring Only
Number analyzed (Participants) | 17 | 21 | 19 | 18
standard drinks per person | 22.1 (25.5) | 17.9 (14.9) | 28.1 (50.4) | 23.9 (22.8)

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up (approximately 2 months)
Description: There are no adverse events to report.
Arm/Group | Episodic Future Thinking (EFT) | Volitional Choice (VC) | Episodic Future Thinking Plus Volitional Choice | Monitoring Only
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/21 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/21 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/21 | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT05235971/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT05235971/ICF_000.pdf